CLINICAL TRIAL: NCT03567525
Title: The Effect of a Peritoneal Iliac Flap on Lymphocele Formation After Robotic Radical Prostatectomy
Brief Title: Peritoneal Iliac Flap and Lymphocele Formation After Robotic Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HHC-2018-0115
Record Dates: First submitted 2018-06-13; First posted 2018-06-25 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Lymphocele After Surgical Procedure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Neither the patient nor the surgeon (who is also the investigator) will know to which arm patients are randomized (standard surgical approach) or experimental approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard surgical approach (Active Comparator): standard lymphadenectomy using clips and bipolar cautery to seal lymphatic vessels
  Interventions: Procedure: Standard surgical approach
- Experimental approach (Experimental): lymph node dissection using the peritoneal iliac flap approach to seal lymphatic vessels
  Interventions: Procedure: lymph node dissection using the peritoneal iliac flap approach to seal lymphatic vessels

INTERVENTIONS:
Procedure: lymph node dissection using the peritoneal iliac flap approach to seal lymphatic vessels — After pelvic lymph node dissection, lymphatic vessels will be sealed by formation of a peritoneal iliac flap in which the bladder in folded over the area of lymph node dissection
  Arms: Experimental approach
Procedure: Standard surgical approach — After pelvic lymph node dissection, lymphatic vessels will be sealed using the standard approach
  Arms: Standard surgical approach

SUMMARY:
Lymphoceles are a potentially serious complication of radical prostatectomy (RP) with pelvic lymph node dissection. They are associated with abdominal pain, urinary tract symptoms, fever, lower extremity swelling and deep vein thrombosis. They can be severe enough to necessitate intervention in 5% of patients after RRP with PLND, with sequela that could include infection and nerve damage. Studies evaluating strategies to preclude lymphocele formation after RP have included comparisons of the use of titanium clips vs bipolar coagulation to seal lymphatic vessels during pelvic lymph node dissection. In a recent prospective randomized trial comparing these approaches, no differences were observed in the rates of lymphocele formation as detected by ultrasound. There is a need to continue to test potential strategies to minimize the formation of lymphoceles after RRP.

Creation of a peritoneal iliac flap is one approach has potential towards this end. At the Lahey Hospital and Medical Center in Burlington, MA surgeons routinely fold the bladder into a peritoneal flap to overlay the area of extended lymphadenectomy. It is thought that this method prevents the formation of lymphoceles because the flap creates a window, which allows drainage of the lymph fluid into the peritoneal cavity to be reabsorbed. While the Lahey study supports the safety and effectiveness of the peritoneal flap approach, the procedure has never been evaluated through a randomized prospective trial and the practice is certainly not standard of care. We therefore propose a randomized, prospective clinical trial to be conducted in the Hartford Hospital Urology Department to examine the effectiveness of a peritoneal iliac flap on the formation of lymphoceles after RRP with pelvic lymph node dissection.

Hypotheses:

1. We hypothesize that, at 3 months after RP, rates of lymphocele formation (symptomatic and asymptomatic lymphoceles) will be significantly lower in patients who have pelvic lymph node dissection using the peritoneal iliac flap approach than in patients who have pelvic lymph node dissection using the standard approach.
2. Lymphoceles are often associated with lower urinary tract symptoms. We hypothesize that, after RP, severity of urinary bother symptoms and urinary incontinence will be significantly lower at each measurement period for patients who had pelvic lymph node dissection using the peritoneal iliac flap approach relative to patients who had pelvic lymph node dissection using the standard approach.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo robotic assisted radical prostatectomy with pelvic lymph node dissection for prostate cancer at Hartford Hospital.
* diagnosed with biopsy-proven prostate cancer, with intermediate or high risk features per D'Amico risk stratification
* ability to give informed consent to participate in the study

Exclusion Criteria:

* Patients with prior prostate irradiation and peri-aortic lymph node dissections will be excluded

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Lymphocele formation | 3 months
  Formation of a least one lymphocele as detected by pelvic ultrasound 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No